CLINICAL TRIAL: NCT02642068
Title: Neuropsychology, Neuroimage and Neurophysiology in Adults With Attention-Deficit Hyperactivity Disorder: An Endophenotype and Follow-up Study
Brief Title: Neuropsychology, Neuroimage and Neurophysiology in Adults With ADHD
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201401024RINC
Record Dates: First submitted 2014-08-25; First posted 2015-12-30 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Drug-naïve Adult ADHD; Neuropsychology; Neurophysiology; Neuroimaging; Follow-up
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The subjects will receive blood withdrawal. The blood sample will be used for establishing lymphoblastoid cell lines, which will be used for molecular genetic experiments
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- ADHD group: Drug-naïve adult ADHD Probands
- Sibling group: Unaffected Siblings of Drug-naïve Adult ADHD
- Control group: Age-, sex-, handedness-, and IQ-matched controls without lifetime ADHD or a family history of ADHD

SUMMARY:
We anticipate that drug-naïve ADHD probands, particularly those with DAT1 or SLC6A2 gene variants may have higher level of altered microstructural integrity of frontostriatal (FS), frontoparietal (FP), other hypothesized fiber tracts and decreased brain activity of FS, FP, and other circuits, deficits in ERP, and impaired EF, SA, IIA and VM than probands without DAT1 or SLC6A2 gene variants or adult neurotypical. The alterations in the structural and functional connectivity, neurophysiological and neuropsychological functioning would be observed in the unaffected siblings as compared to neurotypical. The unaffected siblings will be in the intermediate position between drug-naïve adult ADHD probands and neurotypical. The genetic dosage is anticipated to pose the strongest effects on the cortical thickness, brain volume, gyrification and microstructural property of white matter, followed by neurophysiology, functional connectivity, and neuropsychological function with the least effect.

In terms of longitudinal follow-up part, we also anticipated despite increasing thinning of cortical thickness, microstructural integrity of several targets fiber tracts, and brain activity of target brain regions and improving performance in EF, SA, IIV, VM from childhood to late adolescence and young adulthood in the neurotypical group, the slopes of developmental trajectories of these neuroimaging and neuropsychological function are lower in the ADHD group.

DETAILED DESCRIPTION:
Attention deficit/hyperactivity disorder (ADHD) is a common (3-10%), early-onset, clinically and genetically heterogeneous neuropsychiatric disorder with lifelong neuropsychological deficits. Despite extensive research in adult ADHD in western countries, there has been no published data about adult ADHD in Taiwan except the PI's and colleagues' previous works on pharmacotherapy in adults with ADHD and only few endophenotype studies based on adults with ADHD in the world. The ultimate goals of this 5-year project are to identify which neuropsychological, functional and structural connectivity, and neurophysiological variables can be effective endophenotypes (biomarkers) for ADHD based on unaffected sibling (1st-3rd years) and follow-up (4th-5th years) designs. With the accomplishment of the following study goals, this study will be the first study on the topics of neuroimaging and neurophysiological endophenotypes on adult ADHD using advanced imaging techniques (i.e., Tract-based autonomic analysis, TBAA) and comprehensive clinical and neurocognitive data. This proposal has one primary aim and four secondary aims:

Primary Aim:

1. To validate structural (assessed by TBAA using diffusing spectrum imaging, DSI) and functional connectivity (assessed by resting-state fMRI) in frontostriatal, frontoparietal and other circuitries, and neurophysiological functions (assessed by stop-signal event-related potential [ERP]: N2, P3, ERN, Pe) as effective imaging endophenotypes by demonstrating the intermediate position of unaffected siblings between ADHD probands, and age-, sex-, handedness-, and IQ-matched adult neurotypical and association with DAT1 and NET (SLC6A2) variants;

   Secondary Aims:
2. To validate the executive functions (EF), sustained attention (SA), intraindividual variability (IIV), visual-spatial memory (VM) as effective neurocognitive endophenotypes by demonstrating the intermediate position of unaffected siblings between ADHD probands, and adult neurotypical;
3. To examine the developmental trajectory and stability of neuropsychological functions and structural and functional connectivity from childhood to adolescence and young adulthood;
4. To correlate the data from structural (morphometric, cortical thickness, gyrification, fiber tract integrity) and functional connectivity (rsfMRI), neuropsychology (Executive function, visual-spatial memory, sustained attention, variability), neurophysiology (Stop-signal ERP) and ADHD core symptoms stratifying by the presence of ADHD, presence of DAT1 and NET (SLC6A2) variants, proband-unaffected sibling dyads, and different developmental stages.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 16-30, who have clinical diagnosis of a ADHD according to the DSM-IV and DSM-5 diagnostic criteria, and who have never been treated with medication for ADHD treatment. At least 30 out of 60 subjects have same-sex unaffected siblings.

Exclusion Criteria:

* The subjects will be excluded from the study if they meet any of the following criteria: (1) Comorbidity with DSM-IV-TR or DSM-5 diagnoses of autism spectrum disorder, schizophrenia, schizoaffective disorder, delusional disorder, other psychotic disorder, organic psychosis, schizotypal personality disorder, bipolar disorder, depression, severe anxiety disorders or substance use; (2) With neurodegenerative disorder, epilepsy, involuntary movement disorder, congenital metabolic disorder, brain tumor, history of severe head trauma, and history of craniotomy; (3)With visual or hearing impairments, or motor disability which may influence the process of MRI assessment; and (4) Full-scale IQ lower than 80.

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This 5-year proposal consists of two parts: (1) a 3-year case-control study with unaffected siblings and adult neurotypicals as controls to investigate the brain structural connectivity, functional connectivity, neurophysiological, neuropsychological functioning in 60 probands with ADHD, their unaffected siblings (at least 30 same-sex siblings, n=30~60) and age-, sex-, handedness-, and IQ-matched neurotypicals (n=90~120) with estimated total sample size as at least 180 up to 240. (2) a 2-year follow-up study to repeat the neuropsychological and MRI assessments and to assess electrophysiology related to inhibition controls of 40 adolescents and young adults with childhood diagnosis of ADHD and 40 neurotypicals who had same neuropsychological and imaging assessments in 2010.8-1013.7.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Structural neuroimaging | 1 day
  Using diffusing spectrum imaging (DSI) to assess the structural connectivity in frontostriatal, frontoparietal and other circuitries

SECONDARY OUTCOMES:
Functional connectivity of the brain circuits | 1 day
  Using resting-state functional MRI (rsfMRI) to assess the functional connectivity in frontostriatal, frontoparietal and other circuitries.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lee CY, Goh JOS, Gau SS. Differential neural processing of value during decision-making in adults with attention-deficit/hyperactivity disorder and healthy controls. J Psychiatry Neurosci. 2023 Mar 29;48(2):E115-E124. doi: 10.1503/jpn.220123. Print 2023 Mar-Apr. PMID 36990469